CLINICAL TRIAL: NCT05448313
Title: Collaborate2Lose: Collaborating With Romantic and Non-romantic Support Persons to Improve Long-term Weight Loss
Brief Title: Collaborate2Lose: Involving Support Persons in Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 21-101
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: weight loss; body weight changes; body weight
MeSH Terms: conditions — Obesity; Weight Loss; Body Weight Changes; Body Weight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dyadic intervention (Experimental): Veterans and their support person will participate in MOVE!
  Interventions: Behavioral: Dyadic intervention
- Veteran-only intervention (Active Comparator): Veterans will participate in MOVE! alone
  Interventions: Behavioral: Veteran-only intervention

INTERVENTIONS:
Behavioral: Dyadic intervention — Dyads comprising a Veteran and cohabitating support person will participate in the 16-week VA MOVE! weight loss program delivered by video platform. They will then participate in 6 group sessions focused on weight maintenance skills. Communication skills will be taught throughout the intervention.
  Arms: Dyadic intervention
Behavioral: Veteran-only intervention — Veterans will participate in a 72-week weight management program delivered by video platform. 16 sessions will address weight loss, with 6 additional ones addressing weight loss maintenance.
  Arms: Veteran-only intervention

SUMMARY:
This study involves an evaluation of whether social support from a cohabitating adult improves Veteran weight loss in a weight management program.

DETAILED DESCRIPTION:
Dyads comprising a Veteran with obesity and a cohabitating adult will be randomized to participate in a weight management program by the Veteran alone or with their support person. The program will be delivered by research staff using a secure video platform. Outcomes will be assessed remotely at baseline and weeks 24, 48, and 72, with 72 weeks as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria

* aged 18 years or older
* BMI >= 30 kg/m2
* at least one visit with a VA primary care provider within the past year
* weight <=420 lb due to study scale limits
* have been cohabitating and have daily contact over the past 6 months with an adult who can provide support (e.g., spouse/domestic partner, sibling, adult child, friend, family member) for the next 18 months
* desire to lose weight
* able to stand for weight measurements without assistance
* < 2 errors on a validated 6-item cognitive screener
* ability to speak English
* agrees to attend visits per protocol
* individual email-address
* access to hardware and internet connection to enable participation with approved virtual platform Partner inclusion criteria
* aged 18 years or older
* willing to participate
* < 2 errors on a validated 6-item cognitive screener
* ability to speak English
* individual email address

Exclusion Criteria:

Patient exclusion criteria

* active dementia or substance abuse
* history of bariatric surgery or planning to have bariatric surgery in the next 18 months
* pregnancy or planning to become pregnant in the next 18 months, or breastfeeding
* weight loss >= 10 lb in the month prior to screening
* living in a facility such as a nursing home, skilled nursing facility, or assisted living facility
* unable to control what food is purchased and / or served
* impaired hearing
* current use of weight loss medications
* chronic or unstable illness that would limit ability to participate (e.g., recent hospitalization)
* participation in VA MOVE! weight management program in the past 6 months
* current participation in a research or clinical program focusing on lifestyle change
* vomits once or more per week Partner exclusion criteria
* BMI < 18.5 kg/m2
* active dementia or substance abuse
* impaired hearing
* chronic or unstable illness that would impair their ability to provide support
* living in a facility such as a nursing home, skilled nursing facility, or assisted living facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Body weight (lb) | 72 weeks
  Measured on a calibrated, digital scale to the nearest 0.1 lb, assessed every 24 weeks with 72 weeks as the primary endpoint

SECONDARY OUTCOMES:
obesity-specific quality of life | 72 weeks
  Measured on the 31-item, reliable, valid Impact of Weight on Quality of Life-Lite scale. Items are rated on a 5-point graded response scale ranging from never true to always true. Possible scores range from 31 to 155, with greater scores corresponding to greater impairment in quality of life. The measure will be administered every 24 weeks with 72 weeks as the primary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Corrine I. Voils, PhD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT05448313/ICF_000.pdf